CLINICAL TRIAL: NCT05569057
Title: A Phase I Trial of SIM1811-03 in Subjects With Advanced Solid Tumors and Cutaneous T-cell Lymphoma
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jiangsu Simcere Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SIM1811-03-TNFR2-102
Record Dates: First submitted 2022-09-27; First posted 2022-10-06 (Actual); Last update posted 2022-10-07 (Actual); Status verified 2022-10

CONDITIONS: Advanced Solid Tumor; Cutaneous T-cell Lymphoma (CTCL)
MeSH Terms: conditions — Lymphoma, T-Cell, Cutaneous

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- SIM1811-03 Monotherapy (Experimental): All participants receive SIM1811-03 alone
  Interventions: Drug: SIM1811-03

INTERVENTIONS:
Drug: SIM1811-03 — SIM1811-03 is a first-in-class igG-1 based humanized anti-tumor necrosis factor type 2 receptor (TNFR2) monoclonal antibody for the treatment of malignant tumors
  Other Names: SIM0235, TNFR2 monoclonal antibody

SUMMARY:
This is a first in human, open-label, dose escalation and expansion Phase 1 study of SIM1811-03 in adult patients with advanced solid tumors and cutaneous T-cell lymphoma. SIM1811-03 is a first-in-class IgG1-based humanized anti-tumor necrosis factor type 2 receptor (TNFR2) monoclonal antibody for the treatment of malignant tumors.

DETAILED DESCRIPTION:
This is a phase I trial to evaluate the safety, efficacy, and pharmacokinetic/ pharmacodynamic characteristics of SIM1811-03 in subjects with advanced solid tumors and subjects with CTCL.

The trial is composed of two parts, phase Ia and phase Ib. Phase Ia is a dose escalation part to determine the MTD and/or RD of SIM1811-03. Phase Ib is a dose expansion part at RD level SIM1811-03 determined in phase Ia to primarily assess the anti-tumor activity of SIM1811-03 in subjects with solid tumors or CTCL. The tumor types in PhIb will be adjusted based on the response observed in PhIa. Approximately 50 subjects will be enrolled in this phase.

Cohort 1: Patients with CTCL (approximately 20 patients). Cohort 2: Patients with advanced/metastatic solid tumors, including ovarian cancer (approximately 10 patients), NSCLC (approximately 10 patients), and hepatocellular carcinoma etc.

Each subject will undergo Screening, Treatment, Safety Follow-up, and survival Follow-up periods. Any subject who has discontinued from study treatment other than disease progression will also enter PFS follow up period and to continue to have tumor assessments until disease progression, initiation of subsequent anticancer therapies, or death, whichever occurs first. Upon completion of the safety follow up and PFS follow-up, as applicable, all patients, except those who died, withdrew consent or were lost to follow-up, will be followed for survival.

Eligible subjects will receive intravenous infusion of SIM1811-03 on Days 1 and 15 of each 28-day cycle.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent must be obtained prior to any procedures that are not considered standard of care
* ≥18 years old on the day of signing informed consent, male or female
* Histologically and/or cytologically documented advanced/metastatic solid tumors or histologically confirmed CTCL. Patients with lymphoma other than CTCL are not eligible.
* Have relapsed or refractory advanced solid tumors or CTCL, whose disease has progressed during or after standard therapy
* At least one measurable tumor lesion (RECIST 1.1) for patients with solid tumors. Tumor lesions previously treated with radiotherapy or local therapy should not be considered as measurable unless progression is documented.
* For patients with CTCL, the following criteria must be met:

  * Have at least one measurable lesion (mSWAT criteria) , the lesion that has previously been treated with local therapy should not be considered as measurable unless progression is documented;
  * Provide tissue from a punch biopsy of the skin at screening (except for patients in phase Ia dose escalation phase, for whom skin biopsies is recommended only).
  * Mycosis fungoides (MF) or Sézary Syndrome (SS) (Stage IIb-IV based on Tumor Node Metastasis Blood [TNMB] staging system for SS and MF diagnosed at screening) failed of at least 2 prior systemic therapies
  * Meet clinical criteria for systemic treatment (patients that can be treated with radiotherapy and/or skin-directly therapies only are to be excluded)
  * No current large cell transformation
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) of 0 or 1
* Life expectancy of ≥ 12 weeks
* Adequate organ and marrow functions
* Provide archival tumor samples or fresh tumor biopsy (mandatory for Phase Ib, and recommended for Phase Ia)
* Females of childbearing potential require strict contraception during the study

Exclusion Criteria:

* Participated in an interventional clinical trial or has used investigational devices within 28 days prior to first dose of study drug or received any following systemic anti-cancer treatments:

  1. cytotoxic chemotherapy, targeted therapy, immune checkpoint inhibitor within 4 weeks (such as PD-1 inhibitor, PD-L1 inhibitor, or CTLA-4 inhibitor);
  2. radiotherapy within 2 weeks (palliative radiotherapy is allowed at least 1 week before the study drug treatment).
* Toxicity and side effects (due to previous anticancer treatments) have not recovered to ≤ grade 1, unless such AE is not considered to pose safety risks (such as hair loss and neuropathy ≤ grade 2 caused by chemotherapy).
* Required use of corticosteroids for more than 7 consecutive days within 14 days prior to the first dose of study treatment (> 10 mg daily prednisone equivalent for solid tumors; > 20 mg daily prednisone equivalent for CTCL)
* Patients with active or history of or risk of autoimmune disease
* Major surgery (except biopsy) or unhealed wound within 4 weeks prior to first dose of study drug
* Any other current or previous malignancy within the past 2 years except a) adequately treated basal cell or squamous cell skin cancer, b) carcinoma in situ of the cervix, c) carcinoma in situ of the breast d) local prostate cancer after radical resection and/ or definitive radiotherapy with stable prostate specific antigen (PSA) levels for 1 years
* Has known active central nervous system (CNS) metastases
* History of interstitial lung disease, drug-induced interstitial lung disease, radiation pneumonitis, symptomatic interstitial lung disease or evidence of active pneumonia that is not considered appropriate by the investigator
* History of immunodeficiency (including HIV infection)
* Known active hepatitis B or C infection
* Patients with clinically significant cardiovascular diseases
* History of severe allergic reaction to the study drug or excipients used in the protocol
* Has had an allogeneic tissue/solid organ transplant or graft-versus-host disease
* Other conditions that researchers consider inappropriate for inclusion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-09-30 (Estimated); Primary Completion 2024-06-01 (Estimated); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
Phase 1a: Incidence Rate of Dose-Limiting Toxicity (DLT) | Within 28 days after the first dose
  To estimate the maximum tolerated dose (MTD) or recommended dose (RD) of SIM1811-03
Phase 1b: ORR Solid tumors: objective response rate (ORR) assessed by Investigator per RECIST 1.1 CTCL: ORR assessed by Investigator per global response (Olsen 2011) | Assessed up to an average of 1 year
  Phase 1b (dose expansion): To evaluate the anti-tumor activity of SIM1811-03 at the proposed RD

SECONDARY OUTCOMES:
Incidence and severity of adverse events (AEs) | All AEs/SAEs will be collected in this study from the time the subject signs the informed consent form until 90 days after the last dose
  Number of participants with treatment-related adverse events as assessed by CTCAE v5.0".
Incidence of dose interruptions, delays and discontinuations | All AEs/SAEs will be collected in this study from the time the subject signs the informed consent form until 90 days after the last dose
  To assess the tolerability of SIM1811-03
AUC | Days 1, 2, 4, 8, and 15 of Cycle 1 (each cycle is 28 days), then assessed in subsequent cycles, up to an average of 1 year
  To evaluate the area under the curve (AUC) plasma-concentration of SIM1811-03
Cmax | Days 1, 2, 4, 8, and 15 of Cycle 1 (each cycle is 28 days), then assessed in subsequent cycles, up to an average of 1 year
  To evaluate the maximum observed concentration (Cmax) of SIM1811-03 in the blood after a dose is given
Ctrough | Days 1, 2, 4, 8, and 15 of Cycle 1 (each cycle is 28 days), then assessed in subsequent cycles, up to an average of 1 year
  To evaluate the lowest concentration of a drug just before the next dose of SIM1811-03
Tmax | Days 1, 2, 4, 8, and 15 of Cycle 1 (each cycle is 28 days), then assessed in subsequent cycles, up to an average of 1 year
  To evaluate the time take to reach Cmax of SIM1811-03
Half-life (T1/2) | Days 1, 2, 4, 8, and 15 of Cycle 1 (each cycle is 28 days), then assessed in subsequent cycles, up to an average of 1 year
  To evaluate the time it takes for the concentration of SIM1811-03 in the plasma or the total amount in the body to be reduced by 50%
Incidence of anti-drug antibodies (ADAs) to SIM1811-03 | Days 1, 2, 4, 8, and 15 of Cycle 1 (each cycle is 28 days), then assessed in subsequent cycles, up to an average of 1 year
  To assess the occurrence of anti-drug antibodies (ADAs) to SIM1811-03
Titer of anti-drug antibodies (ADAs) to SIM1811-03 | Days 1, 2, 4, 8, and 15 of Cycle 1 (each cycle is 28 days), then assessed in subsequent cycles, up to an average of 1 year
  To evaluate the quasi-quantitative expression of the level of ADA
Overall Response Rate (ORR) | Assessed up to an average of 1 year
  ORR is defined as the proportion of participants who have a partial response (PR) or better per RECIST 1.1
Duration of Response (DOR) | Assessed up to an average of 1 year
  DOR is defined as time from date of initial documentation of a response (PR or better) to date of first documented evidence of PD per RECIST 1.1
Disease Control Rate (DCR) | Assessed up to an average of 1 year
  Disease Control Rate (DCR) is defined as the percentage of patients with advanced or metastatic cancer who have achieved complete response, partial response and stable disease to a therapeutic intervention in clinical trials of anticancer agents
Progression-Free Survival (PFS) | From date of enrollment until the date of first documented progression or date of death from any cause, whichever came first, assessed up to an average of 1 year
  PFS is defined as time from date of first dose of study drug to date of first documented PD, per RACIST 1.1, or death due to any cause, whichever occurs first.
Overall survival (OS) | Up to an average of 2 year
  Overall survival is defined as the duration from the date of enrollment to the date of the participant's death

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - Henry Ford Health, Detroit, Michigan
  - NYU Lagone Health, New York, New York
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Carolina Biooncology Institute, Huntersville, North Carolina
  - Mary Crowley Cancer Research, Dallas, Texas
  - The University of Texas MD Anderson Cancer Center, Houston, Texas